CLINICAL TRIAL: NCT03614949
Title: Phase II Study of Stereotactic Body Radiation Therapy and Atezolizumab in the Management of Recurrent, Persistent, or Metastatic Cervical Cancer
Brief Title: SBRT and Atezolizumab in the Management of Recurrent, Persistent, or Metastatic Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19662; ML40521 (Other: Genentech)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancer; Cervical Cancer Recurrent; Cervical Cancer Metastatic
Keywords: persistent cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiosurgery; Radiotherapy; atezolizumab; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): Stereotactic body radiation therapy (SBRT) followed by atezolizumab, 1 week later.
  Interventions: Radiation: Stereotactic body radiation therapy (SBRT); Drug: Atezolizumab

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy (SBRT) — SBRT with 24 Gy in 3 fractions to participants with ≥ 2 metastatic sites.
  Other Names: radiotherapy
Drug: Atezolizumab — Atezolizumab 1200 mg intravenously (IV) every 3 weeks.
  Other Names: Tecentriq®; immunotherapy

SUMMARY:
The purpose of this study is to see if treatment with atezolizumab and stereotactic body radiation therapy (SBRT) will improve the objective response rate (ORR) compared with atezolizumab alone in patients with recurrent, persistent, or metastatic cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Eastern Cooperative Oncology Group (ECOG) ≤ 2 or Karnofsky Performance Status of ≥ 60
* Participants must have recurrent, persistent, or metastatic cervical cancer, including squamous cell, adenocarcinoma, and adenosquamous histologies recurrent, persistent, or metastatic p16+ cell cancer of the vagina or vulva
* Measurable disease per irRECIST

  * Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that site since radiation
  * Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥10 mm (≥1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam.
* Must have at least 2 distinct lesions as documented by imaging studies within 4 weeks prior to randomization
* Consent to biopsy of metastatic site or consent to retrieval of archival tissue

Exclusion Criteria:

* Patients with known brain metastasis
* Active autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, autoimmune thyroid disease, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study
  * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
* History of prior malignancy within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS of > 90%), such as but not limited to, non-melanoma skin carcinoma, ductal carcinoma in situ, or stage I endometrioid uterine cancer, and others at the discretion of the Principal Investigator (PI)
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (TNF)-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy)
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 5 years
  ORR by Immune-Modified Response Evaluation Criteria in Solid Tumors (irRECIST) criteria of SBRT and atezolizumab in the management of recurrent/persistent/metastatic cervical cancer. Complete Response (CR): Disappearance of all lesions; Partial Response (PR): ≥30% decrease in tumor burden, a in the absence of CR; Progressive Disease (PD): ≥20% increase in tumor burden; Stable Disease (SD): Neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to 5 years
  PFS following combined modality management with SBRT and atezolizumab in the management of recurrent/persistent/metastatic cervical cancer. PFS: Time from the date of start of treatment to the investigator-determined date of progression (determined by irRECIST criteria) or death due to any cause, whichever occurs first. Progressive Disease (PD): ≥20% increase in tumor burden
Overall Survival (OS) | Up to 5 years
  OS following combined modality management with SBRT and atezolizumab in the management of recurrent/persistent/metastatic cervical cancer. OS: Time from the date of start of treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Ahmed, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Ohio State University - OSUMC - Wexner Medical Center, Hilliard, Ohio